CLINICAL TRIAL: NCT01457911
Title: A Multicenter, Randomized, Open-label, 2-arm Parallel Group, 20-week Study Comparing the Efficacy and Safety of Fixed-dose Combination of 1 mg Glimepiride and 250 mg Metformin (AMARYL M 1/250 mg) Versus Glimepiride (AMARYL®) in Chinese Type 2 Diabetes Patients Inadequately Controlled With Metformin.
Brief Title: Evaluation of Fixed Dose Combination of Glimepiride and Metformin in Chinese Type 2 Diabetes Patients Inadequately Controlled With Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC11761; U1111-1121-6792 (Other: UTN)
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMARYL M (Glimepiride and Metformin hydrochloride combination) (Experimental): AMARYL M at a dosage regimen from 1 tablet to 6 tablets, once during a meal or twice during a meal
  Interventions: Drug: Glimepiride and Metformin hydrochloride combination (HOE490)
- AMARYL (Glimepiride) (Active Comparator): AMARYL at a dosage regimen from 1 mg to 6 mg, once during a meal or twice during a meal
  Interventions: Drug: Glimepiride (HOE490)

INTERVENTIONS:
Drug: Glimepiride and Metformin hydrochloride combination (HOE490) — Pharmaceutical form:tablet Route of administration: oral
  Arms: AMARYL M (Glimepiride and Metformin hydrochloride combination)
Drug: Glimepiride (HOE490) — Pharmaceutical form:tablet Route of administration: oral
  Arms: AMARYL (Glimepiride)

SUMMARY:
Primary Objective:

* To evaluate the efficacy of fixed dose combination of glimepiride and metformin (AMARYL M 1/250mg) in comparison with glimepiride (AMARYL) alone in terms of glycemic control as reflected by HbA1c during a 20-week treatment period in patients with type 2 diabetes mellitus (T2DM) inadequately controlled with metformin.

Secondary Objectives:

* To evaluate the percentage of patients reaching HbA1c < 7% or HbA1c ≤ 6.5% of fixed dose combination of 1 mg glimepiride and 250 mg metformin (AMARYL M 1/250mg) in comparison with glimepiride (AMARYL) alone at week 20.
* To evaluate the effect on Fasting Plasma Glucose of fixed dose combination of glimepiride and metformin (AMARYL M 1/250mg) in comparison with glimepiride (AMARYL) alone at week 20.
* To assess the safety and tolerability of fixed dose combination of glimepiride and metformin (AMARYL M 1/250mg).

DETAILED DESCRIPTION:
The study consists of an up to 2-week screening period, a 20-week treatment period, and a 3-day safety follow-up period. Total study duration is up to 23 weeks.

ELIGIBILITY:
Inclusion criteria:

* Chinese patients with type 2 diabetes mellitus, as defined by World Health Organization, diagnosed for at least 1 year at the time of screening visit and inadequately controlled with metformin
* Signed written informed consent

Exclusion criteria:

* Type 1 diabetes mellitus
* HbA1c < 7% or > 10%
* Fasting plasma glucose > 250 mg/dL (> 13.9 mmol/L)
* Age <18 years or Age ≥ 80 years
* Patients who have not been on stable daily dose of at least 1500 mg metformin within 3 months prior to screening
* Patients currently receiving or who have received anti-diabetic drugs other than metformin within 3 months prior to screening

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Absolute change in HbA1c | 20 weeks, from baseline to week 20

SECONDARY OUTCOMES:
Percentage of patients reaching HbA1c < 7% or HbA1c ≤ 6.5%, respectively | 20 weeks, at week 20
Absolute change in Fasting Plasma Glucose | 20 weeks, from baseline to week 20
Number of patients reporting adverse events | 20 weeks, from baseline to week 20
Number of patients reporting serious adverse events | 20 weeks, from baseline to week 20
Hypoglycemia | 20 weeks, from baseline to week 20
Vital signs | 20 weeks, from baseline to week 20
Hematology, Serum chemistry and lipids | 20 weeks, from baseline to week 20

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (22):
- China (22):
  - Investigational Site Number 156001, Beijing
  - Investigational Site Number 156016, Beijing
  - Investigational Site Number 156003, Beijing
  - Investigational Site Number 156018, Beijing
  - Investigational Site Number 156002, Beijing
  - Investigational Site Number 156019, Changchun
  - Investigational Site Number 156017, Chengdu
  - Investigational Site Number 156014, Guangzhou
  - Investigational Site Number 156022, Guangzhou
  - Investigational Site Number 156011, Hangzhou
  - Investigational Site Number 156012, Hefei
  - Investigational Site Number 156020, Jinan
  - Investigational Site Number 156023, Jinan
  - Investigational Site Number 156010, Shanghai
  - Investigational Site Number 156006, Shanghai
  - Investigational Site Number 156009, Shanghai
  - Investigational Site Number 156021, Shenyang
  - Investigational Site Number 156005, Shijiazhuang
  - Investigational Site Number 156004, Taiyuan
  - Investigational Site Number 156024, Tianjin
  - Investigational Site Number 156008, Wuhan
  - Investigational Site Number 156015, Xiamen